CLINICAL TRIAL: NCT00133263
Title: Effectiveness of "Primary Bereavement Care" (PBC) in Widows: A Cluster Randomized Controlled Trial
Brief Title: Effectiveness of a Standardized Bereavement Intervention in Primary Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carlos III Health Institute (Other Government)
Collaborators: Health Department of the Basque Government (Unknown)
Responsible Party: Jesus Angel García García, Basque Health Service / Osakidetza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI020827; 200011007
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2008-03

CONDITIONS: Bereavement; Grief
Keywords: Randomized controlled trial; Primary Care
MeSH Terms: interventions — Primary Health Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Primary Bereavement Care
- 2 (Active Comparator)
  Interventions: Behavioral: the current bereavement care in primary care

INTERVENTIONS:
Behavioral: Primary Bereavement Care — a standardized bereavement intervention in Primary Care
  Other Names: Bereavement Primary Care; Bereavement Intervention in Primary Care; Grief Intervention in Primary Care
  Arms: 1
Behavioral: the current bereavement care in primary care — the non-standardized bereavement care that usually provided family physicians in primary care
  Other Names: The current grief care in primary care
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy of "Primary Bereavement Care" (PBC) -a standardized bereavement intervention- delivered by family physicians (FP), in widows.

DETAILED DESCRIPTION:
Nowadays there is little evidence about what is the best bereavement intervention in primary care and each family physician (FP) assists bereaved people in a different way. The death of a loved one is the most stressful life event that can face a person; in fact, bereavement is associated with an increased risk of depression, generalized anxiety and panic disorder, alcohol abuse and use of medications, sudden cardiac events, suicide, and an increased demand for health resources. The FP is the only specialist who -through his position in the health system and in the community- can give emotional support to the bereaved and simultaneously deal with the health problems associated with the process. In response to this, our work group has designed a guide specifically for FP: Primary Bereavement Care (PBC), and is currently testing its efficacy in a randomized controlled study.

Comparison (s): Recently widows attended by FP trained in PBC through seven PBC sessions, compared to recently widows attended by FP not trained in PBC through seven "ordinary" sessions.

ELIGIBILITY:
Inclusion Criteria:

* Partner death during the last 3 months.

Exclusion Criteria:

* Partner death through suicide or AIDS.
* Son or daughter death during the last 3 years.
* Parent or sibling death the year before.
* Alcohol or drug abuse.
* Psychotic disorder or dementia.
* To be confined to bed
* Illiteracy.

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2001-01; Primary Completion 2005-04 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Texas Revised Inventory of Grief (TRIG) | at 3, 9, 15 and 21 months since death

SECONDARY OUTCOMES:
Grief Experience Inventory (GEI) | at 3, 9, 15 and 21 months since death
General Health Questionnaire - 28 items (GHQ-28) | at 3, 9, 15 and 21 months since death
SF-36 Health Profile (SF-36) | at 3, 9, 15 and 21 months since death

CONTACTS AND LOCATIONS:
Overall Officials: Jesus A. Garcia, MD, Principal Investigator — Primary Care Research Unit of Bizkaia, Basque Health Service/Osakidetza.
Locations (1):
- Primary Care Research Unit of Bizkaia, Basque Health Service/Osakidetza, Bilbao, Bizkaia, Spain

REFERENCES:
- [Background] Garcia Garcia JA, Landa Petralanda V, Trigueros Manzano MC, Gaminde Inda I. [Texas revised inventory of grief: adaptation to Spanish, reliability and validity]. Aten Primaria. 2005 Apr 30;35(7):353-8. doi: 10.1157/13074293. Spanish. PMID 15871796
- [Background] Garcia-Garcia JA, Landa Petralanda V, Trigueros Manzano MC, Gaminde Inda I. [Inventory of experiences in grief (IEG): adaptation to Spanish, reliability and validity]. Aten Primaria. 2001 Feb 15;27(2):86-93. doi: 10.1016/s0212-6567(01)78779-3. Spanish. PMID 11256097
- [Background] Garcia-Garcia JA, Landa Petralanda V, Trigueros Manzano MC, Calvo Aedo P, Gaminde Inda I. [Grief for loss of a spouse: a study with discussion groups in primary care]. Aten Primaria. 1996 Nov 30;18(9):475-9. Spanish. PMID 9280441
- See also: Landa V, García JA. Duelo. Guías Clínicas. Cuidados Primarios de Duelo. 2011. This is a summary in Spanish of the intervention - Primary Bereavement Care - which is used in our project. — https://www.fisterra.com/guias-clinicas/cuidados-primarios-duelo/